CLINICAL TRIAL: NCT01410487
Title: Effects of Weight Loss on Cardio-respiratory Function and Patient-centered Outcomes in an Underserved, Minority Population With Clinically Severe Obesity
Brief Title: Effects of Weight Loss on Cardio-respiratory Function
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 11-01998
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Obesity; Cardiovascular Abnormalities
Keywords: pulmonary circulation
MeSH Terms: conditions — Obesity; Cardiovascular Abnormalities

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese group

SUMMARY:
Obesity is a medical problem of epidemic proportions and is associated with high mortality. Obesity has significant effects on the cardiovascular system, producing structural cardiovascular changes including myocardial hypertrophy, fatty infiltration, and fibrosis; diastolic and systolic dysfunction; changes in pulmonary artery compliance; and increased aortic stiffness - all of which can lead to heart failure. Indeed, evidence suggests that obesity increases the risk for heart disease independent of other known risk factors such as coronary artery disease, hypertension, diabetes mellitus, and obstructive sleep apnea. Obesity also causes significant changes in pulmonary function, including a decrease in expiratory reserve volume and functional residual capacity and closure of peripheral airways. The exact mechanisms for the development of cardiopulmonary disease are not well understood - the pathophysiology is complex and likely multifactorial, related to altered hemodynamic load, altered metabolic activity, underlying inflammation, and increased cardiac output.

Newer diagnostic modalities available at our institution such as cardiac MRI and pulmonary function tests with impulse oscillometry allow us to better evaluate cardiopulmonary dysfunction in patients with severe obesity. Cardiac MRI is especially promising as a non-invasive imaging modality in obese individuals, providing more reproducible measurements of cardiac and vascular anatomy and function relative to echocardiography. Similarly, pulmonary function testing with impulse oscillometry is more sensitive for detection of abnormalities in the distal airways especially when spirometry is normal, as frequently occurs in the severely obese symptomatic patients. The main objective of the proposed study is to evaluate the effect of obesity on quality of life and health care utilization and its relationship to cardiopulmonary disease in an ethnically diverse, underserved obese population by using state-of-the-art diagnostic modalities before and after significant (20%) weight loss.

The investigators propose to perform stress cardiac MRI and pulmonary function testing with oscillometry before and after significant surgical weight loss in 150 severely obese patients with cardiopulmonary symptoms. Patients evaluated in the comprehensive Obesity Center at Bellevue Hospital who meet NIH Consensus Guidelines for Bariatric Surgery, who have cardiopulmonary symptoms, and who meet clinical criteria for cardiac stress testing and pulmonary function testing will be approached by the study personnel and offered enrollment. Informed consent will be obtained. Enrolled patients will undergo clinical evaluation with a detailed medical history including the Borg dyspnea scale, physical examination, laboratory testing including cardiopulmonary biomarkers (brain natriuretic peptide, C-reactive protein, atrial natriuretic peptide), and non-invasive cardiovascular stress MRI and pulmonary physiologic evaluation including spirometry, plethysmography and impulse oscillometry (IOS). Patients with active smoking history and/or asthma will be identified clinically.

Cardiovascular MRI will be performed using a 1.5T (Avanto or Espree, Siemens Healthcare) system. Standard cardiovascular techniques will be used for the assessment of myocardial and vascular structure and function, including T1-weighted, T2-weighted, late gadolinium enhancement, cine, tagged and phase contrast imaging in selected planes. Adenosine stress MRI will be performed for evaluation of underlying coronary artery or microvascular disease.

ELIGIBILITY:
Inclusion Criteria:

Eligible patients for this study are patients who are booked for bariatric surgery and who have cardiopulmonary symptoms that require further cardiopulmonary testing prior to bariatric surgery.

Exclusion Criteria:

Patients with contraindications to MRI examination with gadolinium contrast and adenosine administration will be excluded. Additional exclusions include being deemed unable to comply with the study protocol (either self-selected or by indicating during screening that s/he could not complete all requested tasks), participation in other obesity- or diabetes-related clinical trials, or diagnosis of cognitive dysfunction or significant psychiatric comorbidity.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients utilizing the Bariatric Clinic services at Bellevue (City/Public) Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Effects of body mass & adiposity on airway mechanics and cardiovascular anatomy and physiology. | 2 years
  Detailed evaluation of quality of life, health care utilization and the cardiopulmonary system in severe obesity, with an assessment of the correlation between specific cardiovascular and pulmonary parameters to improve our understanding and treatment of symptomatic obese patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Bellevue Hospital Ambulatory Cinic - Suite 1D, New York, New York, United States